CLINICAL TRIAL: NCT05054829
Title: Establishment of Social Skills Training Group in Adults With Autism Spectrum Disorder and Effectiveness Analysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201612185RINC
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-03

CONDITIONS: Social Skill Training Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEERS (Experimental)
  Interventions: Behavioral: PEERS®: program for the education and enrichment of relational skills
- Controls (Other)
  Interventions: Behavioral: PEERS®: program for the education and enrichment of relational skills

INTERVENTIONS:
Behavioral: PEERS®: program for the education and enrichment of relational skills — providing evidence-based social skills treatment to preschoolers, adolescents, and young adults with autism spectrum disorder (ASD)

SUMMARY:
This project aims to examine the effectiveness of social skill training group in adults with autism spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 45 years
* having relational problems
* having motivation to participate
* good chinese speaking
* having a healthy cargiver join together
* IQ > 70 (WAIS)
* Autism Spectrum Quotient > 26

Exclusion Criteria:

* ever had psychosis and neurological diseases
* visual and hiring impairment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Outcome analysis | after intervention 12 weeks
  Background characteristics, co-existing psychiatric conditions and dropout rates for the two groups are compared using χ2 tests. Differences between two groups' baseline measures are analyzed using two-sided independent t tests.
  The comparison will adopt an intention-to-treat principle. The missing data are substituted with last observation carried forward. To analyze the reasons for the attrition, the dropouts will also be compared to the completers on their clinical variables.
  Then, repeated-measures analyses of variance (ANOVAs) are used to calculate between- and within-group effects on all continuous variables. Treatment effect calculations (Cohen's d) will be calculated for each indicator. Differences between the interventions in CGI-I will be examined using a one-way ANOVA. Reported change in the follow-up survey was compared between the PEERS group and the controls using independent t tests.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided